CLINICAL TRIAL: NCT03446560
Title: Cloud Based Follow up of CPAP Treatment in Sleep Apnea Patients - a Multi Center Randomized Controlled Trial
Brief Title: Cloud Based Follow up of CPAP Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Borås Lasarett (Other); Skaraborgs Hospital (Unknown); NU-Hospital Organization, Sweden (Other)
Responsible Party: Principal Investigator, Ludger Grote, MD, Senior Consultant, Professor, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUREG-663941; 227161 (Registry Identifier: Västra Götalands Regionen Researchweb)
Record Dates: First submitted 2018-01-18; First posted 2018-02-27 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea Syndromes
Keywords: Compliance; Telemedicine; Patient related outcome measures
MeSH Terms: conditions — Sleep Apnea Syndromes; Patient Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, multicenter, parallell group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP, conventional follow up (Active Comparator): Follow up of patients after initiation of treatment according to clinical routine at the study site.
  Interventions: Device: CPAP, conventional follow up
- CPAP, telemedicine based follow up (Active Comparator): Follow up of patients after initiation of treatment according to a telemedicine based routine.
  Interventions: Device: CPAP, telemedicine based follow up

INTERVENTIONS:
Device: CPAP, conventional follow up — Positive airway pressure to splint the airway and to prevent apneas during sleep. Follow up of patients after initiation of treatment according to clinical routine at the study site. Patients are informed to call or visit the sleep center in case of problems with the CPAP device. At 3 months a follow up visit is scheduled at the sleep center. CPAP compliance data will be downloaded and all patients fill in a number of questionaires related to the CPAP treatment effects on sleep apnea symptoms and health related quality of Life. Mask fitting will be tested.
  Arms: CPAP, conventional follow up
Device: CPAP, telemedicine based follow up — Follow up of patients by means of a telemedicine solution for surveillance of CPAP treatment, Compliance with and efficacy of CPAP can be followed up by the sleep center personnel on a regular basis. Patients with low compliance and mask fitting problems will be contacted by phone. At the end of the 3 months period a visit at the sleep center will be scheduled only for patients with low compliance, low treatment efficacy, or high mask leakage. All patients will be asked to fill in a number of questionaires related to CPAP treatment effects on sleep apnea symptoms and health related quality of Life.
  Arms: CPAP, telemedicine based follow up

SUMMARY:
Obstructive sleep apnea (OSA) is treated with a continuous positive airway pressure, so called CPAP. A new technology that enables telemetric monitoring of CPAP therapy. This study randomizes 560 patients to A) conventional follow up procedures or B to a telemedicine based follow up procedure. Main endpoint parameter is CPAP treatment compliance at 3 months after start of treatment.

DETAILED DESCRIPTION:
Background:

Obstructive sleep apnea (OSA) is treated with a continuous positive airway pressure, so called CPAP, during sleep. CPAP startup and follow-up is performed at four sleep clinics in the West Swedish Region (SU / S, SÄS, SkaS, NÄL). Patient volumes are high, waiting times are long and long-term follow-up is inconsistent. A new technology that enables telemetric monitoring of CPAP therapy based on transfer of therapy data to a data cloud has been introduced. Healthcare personnel can identify patients with therapy problems.

Data from minor studies suggest several benefits of this telemedicine solution (increased therapeutic capacity, lower patient and community costs and a time benefit for the sleep medicine unit). Today, the sleep Clinical in the region use different procedures for monitoring CPAP treatment.

Scientific question:

Is telemedicine monitoring of CPAP treatment an adequate solution for follow up in all patients ? Is the additional cost of a telemedicine solution balanced by a better outcome after therapy?

Hypothesis:

Intensive telemedicine monitoring, especially at the start of CPAP therapy, leads to improved CPAP care at the participating sleep units.

Method:

The study randomizes 560 patients (moderate to severe sleep apnea) to different CPAP treatment follow up procedures: A) the current routine of the sleep clinic or B) the new telemedicine solution (1: 1 randomization). The main outcome parameter of the study is the mean CPAP use after 3 months of treatment. Secondary outcome parameters include the reduction of sleep apnea intensity, daytime sleepiness, and patient-related outcome measures (PROM).

Aim:

The aim of the study is to map the pros and cons of a telemedicine solution in CPAP therapy regarding treatment outcomes, patient quality of life and resource utilization at the sleep center.

ELIGIBILITY:
Inclusion Criteria:

* Verified sleep apnea diagnosis according to ICSD II criteria
* Indication for CPAP treatment according to Swedish national guidelines
* Capacity to read and understand the Swedish language
* Willingness to test CPAP treatment

Exclusion Criteria:

* Instable concomitant disease requiring frequent hospitalization
* Alcohol and drug abuse
* Non-availability during the follow up during 3 months (e.g. frequent or long-term travelling)
* Hypoventilation syndrome with PCO2>7kpa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
CPAP treatment compliance at 3 months | 3 months
  Mean nightly use of CPAP treatment (h/night) according to the built in time counter of the CPAP device, between group difference

SECONDARY OUTCOMES:
Reduction of daytime sleepiness | 3 months
  Reduction of the score in the Epworth Sleepiness Scale Score (range 0-24, 0=no sleepiness, 24=very high sleepiness, summary score from 8 different questions about the probability of daytime sleepiness, each question can generate between 0=unlikely and 4=highly likely points), assessment at baseline and at follow up, between group difference
Reduction of the degree of sleep apnea | 3 months
  Between Group difference in the reduction of the Apnea Hypopnea Index (n/h) from baseline (no treatment) to follow up (with CPAP on)
Non Acceptance Rate of CPAP therapy | 3 months
  Proportion of patients refusing CPAP therapy, between group difference
Health care utilization during follow up | 3 months
  Time spent for follow up procedures by the Health care personel, between group difference
Patient satisfaction regarding the follow up procedure | 3 months
  Visual Analogue Scale (VAS) Rating of patient satisfaction with the two different follow up procedures, VAS scale has 0 to 100 Points where 0=very low satisfaction and 100= very high satisfaction, no subscales.

OTHER OUTCOMES:
Degree of comorbid depression and anxiety symptoms | 3 months
  Score of the Hospital Anxiety and Depression Scale (HADS) pre and post treatment, between group differences. The HADS scale consists of 7 questions for anxiety rating (each question can generate 0-1 Point), the points from each question will be summarized to a total score with has a range of 0-21 (0=no anxiety and 21=severe anxiety). The depression rating is performed according to the same principle (seven questions, summary score with a range 0 to 21).
Degree of comorbid insomnia | 3 months
  Score of the Insomnia Severity Index (ISI) Score pre and post treatment, between group differences. The questionnaire consists of 7 questions, each generating 0 (no insomnia problem) or up to 4 (very severe insomnia problems) Points. The 7 questions can generate a summary score between 0 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Grote, Principal Investigator — Respiratory Medicine, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Sleep Disorders Center, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fridriksson B, Berndtson M, Hamnered H, Faeder E, Zou D, Hedner J, Grote L. Beneficial Effects of Early Intervention Telemedicine-based Follow-Up in Sleep Apnea: A Randomized Controlled Multicenter Trial. Ann Am Thorac Soc. 2023 Oct;20(10):1499-1507. doi: 10.1513/AnnalsATS.202208-723OC. PMID 37463309